CLINICAL TRIAL: NCT06884761
Title: The Effect of Routine Activity on the Risk for Preterm Delivery in Women With a Short Cervix. A Randomized Control Trial
Brief Title: Routine Activity and Preterm Delivery Risk in Women With a Short Cervix
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 124-24-WOMC
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cervical Shortening
Keywords: Preterm delivery; Physical activity; cervical shortening; Bed rest; Cervical length; High-risk pregnancy; Randomized controlled trial
MeSH Terms: conditions — Premature Birth; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maximal Rest (Experimental): Participants in this group are instructed to follow maximal rest protocols. They are advised to avoid strenuous activities, including prolonged standing, lifting heavy objects, or engaging in physically demanding tasks. This group represents the traditional bed rest approach to managing pregnancies with a short cervix.
  Interventions: Behavioral: Maximal Rest
- Routine Activity (No Intervention): Participants in this group are encouraged to maintain routine, non-strenuous physical activity. They are not instructed to follow bed rest but are asked to avoid overtly strenuous activities. This group reflects the standard approach of allowing typical daily activity without additional restrictions.

INTERVENTIONS:
Behavioral: Maximal Rest — Participants in this group are instructed to follow maximal rest protocols. They are advised to avoid strenuous activities, including prolonged standing, lifting heavy objects, or engaging in physically demanding tasks. This group represents the traditional bed rest approach to managing pregnancies with a short cervix.
  Arms: Maximal Rest

SUMMARY:
The goal of this clinical trial is to evaluate the effect of routine activity versus rest on the risk of preterm delivery in pregnant women with a short cervix diagnosed between 24 and 34 weeks of gestation. The main questions it aims to answer are:

Does routine activity influence the gestational age at delivery? How does routine activity affect secondary outcomes such as preterm labor, premature rupture of membranes, delivery mode, maternal anxiety, and satisfaction?

Researchers will compare women instructed to maintain routine activity (control group) to women advised to practice maximal rest (intervention group) to see if physical activity impacts preterm birth outcomes.

Participants will:

Wear a smart band to monitor step counts over a two-week period. Be randomized into two groups: one encouraged to maintain routine activity and the other advised to follow strict rest protocols.

Undergo regular follow-ups at a high-risk pregnancy clinic and have their data collected through hospital records and smart band tracking.

This randomized controlled trial will assess gestational age at delivery as the primary outcome, along with secondary maternal and neonatal outcomes, providing insight into the role of physical activity in managing pregnancies complicated by a short cervix.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies between 24+0 and 34+6 weeks.
* Short cervical length (<25 mm) confirmed via transvaginal ultrasound.
* No medical contraindications to physical activity.

Exclusion Criteria:

* Twin pregnancies or higher-order multiples.
* Medical indications for reduced mobility (e.g., symphysiolysis, fall risk).
* Maternal comorbidities, fetal distress, vaginal bleeding, PPROM, or need for immediate delivery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female
Enrollment: 100 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-12-29 (Estimated); Study Completion 2027-12-29 (Estimated)

PRIMARY OUTCOMES:
gestational age at delivery | two years
  to assess the effect of physical activity on the gestational age at delivery.

SECONDARY OUTCOMES:
Rates of preterm labor. | two years
Incidence of premature rupture of membranes (PPROM). | two years
Mod of delivery (cesarean, instrumental, or spontaneous). | two years

CONTACTS AND LOCATIONS:
Locations (1):
- The Edith Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zemet R, Schiff E, Manovitch Z, Cahan T, Yoeli-Ullman R, Brandt B, Hendler I, Dorfman-Margolis L, Yinon Y, Sivan E, Mazaki-Tovi S. Quantitative assessment of physical activity in pregnant women with sonographic short cervix and the risk for preterm delivery: A prospective pilot study. PLoS One. 2018 Jun 11;13(6):e0198949. doi: 10.1371/journal.pone.0198949. eCollection 2018. PMID 29889906
- [Result] Grobman WA, Gilbert SA, Iams JD, Spong CY, Saade G, Mercer BM, Tita ATN, Rouse DJ, Sorokin Y, Leveno KJ, Tolosa JE, Thorp JM, Caritis SN, Peter Van Dorsten J; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network*. Activity restriction among women with a short cervix. Obstet Gynecol. 2013 Jun;121(6):1181-1186. doi: 10.1097/AOG.0b013e3182917529. PMID 23812450
- [Result] Sosa CG, Althabe F, Belizan JM, Bergel E. Bed rest in singleton pregnancies for preventing preterm birth. Cochrane Database Syst Rev. 2015 Mar 30;2015(3):CD003581. doi: 10.1002/14651858.CD003581.pub3. PMID 25821121
- [Result] Teitelman AM, Welch LS, Hellenbrand KG, Bracken MB. Effect of maternal work activity on preterm birth and low birth weight. Am J Epidemiol. 1990 Jan;131(1):104-13. doi: 10.1093/oxfordjournals.aje.a115463. PMID 2293743
- [Result] Maloni JA. Antepartum bed rest for pregnancy complications: efficacy and safety for preventing preterm birth. Biol Res Nurs. 2010 Oct;12(2):106-24. doi: 10.1177/1099800410375978. PMID 20798159
- [Result] Goldenberg RL, Cliver SP, Bronstein J, Cutter GR, Andrews WW, Mennemeyer ST. Bed rest in pregnancy. Obstet Gynecol. 1994 Jul;84(1):131-6. PMID 8008308
- [Result] Berghella V, Saccone G. Cervical assessment by ultrasound for preventing preterm delivery. Cochrane Database Syst Rev. 2019 Sep 25;9(9):CD007235. doi: 10.1002/14651858.CD007235.pub4. PMID 31553800
- [Result] Navathe R, Saccone G, Villani M, Knapp J, Cruz Y, Boelig R, Roman A, Berghella V. Decrease in the incidence of threatened preterm labor after implementation of transvaginal ultrasound cervical length universal screening. J Matern Fetal Neonatal Med. 2019 Jun;32(11):1853-1858. doi: 10.1080/14767058.2017.1421166. Epub 2018 Jan 5. PMID 29303014
- [Result] Blencowe H, Cousens S, Chou D, Oestergaard M, Say L, Moller AB, Kinney M, Lawn J; Born Too Soon Preterm Birth Action Group. Born too soon: the global epidemiology of 15 million preterm births. Reprod Health. 2013;10 Suppl 1(Suppl 1):S2. doi: 10.1186/1742-4755-10-S1-S2. Epub 2013 Nov 15. PMID 24625129
- [Result] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Result] MacDorman MF, Kirmeyer S. Fetal and perinatal mortality, United States, 2005. Natl Vital Stat Rep. 2009 Jan 28;57(8):1-19. PMID 19294965
- [Result] Hamilton BE, Martin JA, Osterman MJ. Births: Preliminary Data for 2015. Natl Vital Stat Rep. 2016 Jun;65(3):1-15. PMID 27309256
- [Result] Society for Maternal-Fetal Medicine Publications Committee, with assistance of Vincenzo Berghella. Progesterone and preterm birth prevention: translating clinical trials data into clinical practice. Am J Obstet Gynecol. 2012 May;206(5):376-86. doi: 10.1016/j.ajog.2012.03.010. PMID 22542113
- [Result] WHO: recommended definitions, terminology and format for statistical tables related to the perinatal period and use of a new certificate for cause of perinatal deaths. Modifications recommended by FIGO as amended October 14, 1976. Acta Obstet Gynecol Scand. 1977;56(3):247-53. No abstract available. PMID 560099

DOCUMENTS (1):
  • Study Protocol (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT06884761/Prot_000.pdf